CLINICAL TRIAL: NCT07396792
Title: Screening for Cardiac and Cardiac-associated Pathology Using Single-channel Electrocardiogram Analyzed With Machine Learning Models
Brief Title: Screening for Cardiac and Cardiac-associated Pathology Using Single-channel Electrocardiogram
Status: Not yet recruiting | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: ChPSH135Pif
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Arterial Hypertension; Heart Rhythm Disorders; Valvular Heart Diseases; Heart Failure; Diabetes Mellitus; Chronic Kidney Disease (Stage 3-4); Metabolic Syndrome; Coronary Artery Disease
Keywords: Screening; Electrocardiogramm; single-channel electrocardiogram; machine learning models; Coronary artery disease; diabetes mellitus; metabolic syndrome; anemia; hypercholesterolemia; arterial hypertension
MeSH Terms: conditions — Hypertension; Arrhythmias, Cardiac; Heart Valve Diseases; Heart Failure; Diabetes Mellitus; Renal Insufficiency, Chronic; Metabolic Syndrome; Coronary Artery Disease; Anemia; Hypercholesterolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training sample: 2500 of patients 18 years old and older with and without cardiac and cardiac-associated pathology confirmed by the results of full examination (laboratory, clinical and instrumental) and by results of the spectral analysis of electrocardiogram (the parameters listed below will be calculated as the median of the tact-cycle: TpTe, VAT, QTc, QT / TQ, QRS_E, T_E, TP_E, BETA, BETA_S, BAD_T, QRS_D1_ons, QRS_D1_offs, QRS_D2, QRS_Ei (i = 1,2,3,4), T_Ei (i= 1,2,3,4), HFQRS, QRSw, RA, SA, TA and others).
- Test sample: 1500 of patients 18 years old and older with and without cardiac and cardiac-associated pathology confirmed by the results of full examination (laboratory, clinical and instrumental) and by results of the spectral analysis of electrocardiogram (the parameters listed below will be calculated as the median of the tact-cycle: TpTe, VAT, QTc, QT / TQ, QRS_E, T_E, TP_E, BETA, BETA_S, BAD_T, QRS_D1_ons, QRS_D1_offs, QRS_D2, QRS_Ei (i = 1,2,3,4), T_Ei (i= 1,2,3,4), HFQRS, QRSw, RA, SA, TA and others).

SUMMARY:
It is a prospective, controlled, single-center, observational, non-randomized study. The study is planned to include at least 4000 patients 18 years old and older in the training sample and 1000 patients over 18 years old in the test sample (the total number of patients is at least 5000 people). Patients will be included in the study if they have undergone a full examination (laboratory, clinical and instrumental), allowing for the verification or exclusion of cardiac and cardiac-associated pathology in accordance with current recommendations. During the course of the study, the authors of the work do not interfere with the above-mentioned scope of the examination, which is carried out on patients in accordance with clinical guidelines. All patients included in the study will undergo ECG recording in standard lead I for 1 minute twice, followed by spectral analysis of the obtained data, which will be stored at the remote monitoring center of Sechenov University without being linked to the personal data of patients. A spectral analysis of the electrocardiogram will be performed using a continuous wavelet transform. The result of this study will be the identification of ECG parameters that will correlate with cardiac and cardiac-associated pathology

DETAILED DESCRIPTION:
The aim of the study: to create, evaluate the diagnostic efficiency and pilot application of a method for screening cardiac and cardiac-associated pathology based on the analysis of a single-channel electrocardiogram using elements of artificial intelligence. It is a prospective, controlled, single-center, observational, non-randomized study. The study is planned to include at least 4000 patients over 18 years old in the training sample and 1000 patients 18 years old and older in the test sample (the total number of patients is at least 5000 people). Patients will be included in the study if they have undergone a full examination (laboratory, clinical and instrumental), allowing for the verification or exclusion of cardiac and cardiac-associated pathology in accordance with current recommendations. To detect heart defects and heart failure: an expert echocardiography protocol, blood tests for cardiac-specific markers, and stress tests if indicated. To detect coronary artery disease: detection of significant coronary stenosis during coronary artery imaging: myocardial perfusion or determination of fractional coronary flow reserve, or stress echocardiography. For hypertension: repeated office blood pressure measurements, 24-hour blood pressure monitoring. For coronary heart disease: resting ECG and long-term Holter monitoring. For cardiac-associated pathology: blood tests: hemoglobin and red blood cell levels, glucose, glycated hemoglobin, oral glucose tolerance test, creatinine, uric acid levels, total cholesterol, low- and high-density lipoproteins, and triglycerides. Additional examination data will be taken into account if performed outside the protocol of this study. During the course of the study, the authors of the work do not interfere with the above-mentioned scope of the examination, which is carried out on patients in accordance with clinical guidelines. All patients included in the study will undergo ECG recording in standard lead I for 1 minute twice, followed by spectral analysis of the obtained data, which will be stored at the remote monitoring center of Sechenov University without being linked to the personal data of patients. Single-channel ECG will be recorded using the portable single-lead ECG monitor CardioQvark. It is designed as an iPhone cover. It is registered with the Federal Service for Health Supervision on February 15, 2019. RZN No. 2019/8124.The patient's personal data (last name, first name, patronymic, date of birth, contact information) will not be transferred or taken into account. Each patient is assigned an individual number that is not associated with his/her personal data. Then a spectral analysis of the electrocardiogram will be performed using a continuous wavelet transform, the principles of which are based on the Fourier transform. The analysis involves the evaluation of the following parameters (the parameters listed below will be calculated as the median of the tact-cycle):• TpTe - time from peak to end of the T-wave• VAT - time from the beginning of the QRS to the R-peak• QTc - corrected QT interval.• QT / TQ - the ratio of QT length to TQ length (from the end of T to the beginning of the QRS of the next complex).• QRS_E - the total energy of the QRS wave based on the wavelet transform• T_E - T-wave total energy based on wavelet transform• TP_E- energy of the main tooth of the T-wave based on the wavelet transform• BETA, BETA_S - T-wave asymmetry coefficients (simple and smooth versions)• BAD_T - flag of T-wave quality (whether expressed in the current lead• QRS_D1_ons - energy of the leading edge of the R-wave (based on the "first derivative" wavelet transform)• QRS_D1_offs - energy of the trailing edge of the R-wave (based on the "first derivative" wavelet transform)• QRS_D2 - peak energy of the R-wave (based on the "second derivative" wavelet transform)• QRS_Ei (i = 1,2,3,4) - QRS-wave energy in 4 frequency ranges (2-4-8-16-32 Hz) based on wavelet transform• T_Ei (i = 1,2,3,4) - T-wave energy in 4 frequency ranges (2-4-6-8-10 Hz) based on wavelet transform• HFQRS - the amplitude of the RF components of the QRS wave. Additionally used parameters:• TpTe, VAT, QTc - are duplicated to control the correctness of the record processing (the value of the UCC should be approximately equal to the median of the tick-by-bar).• QRSw - QRS width.• RA, SA, TA - the amplitudes of the R, S, T-waves, respectively, are used to normalize the parameters listed above.Statistical analysis and modeling will be performed using Python V3.8.8 and R V.4.0, as well as SPSS v.17.The correlation between various combinations of time, amplitude and frequency parameters of ECG and the presence of cardiac and cardiac-associated pathology will be analyzed. Certain parameters will be included in various multivariate analysis models: Lasso regression, Random Forest, Multilayer Perceptron, Support Vector Machine and Decision Tree. The model with the highest diagnostic accuracy will be selected, on which the algorithm will be tested.The outcome of this study will be the development and validation of an algorithm for identifying various cardiac and cardiac-associated pathologies based on the analysis of single-channel ECG parameters. The development of a medical-use program will also be undertaken.Study endpoints: • Single-channel ECG parameters that significantly correlate with the presence of various cardiac and cardiac-related pathologies; • Sensitivity, specificity, and diagnostic accuracy of multivariate models for analyzing single-channel ECG data; • Diagnostic accuracy of the algorithm when tested on a test sample of patients.

ELIGIBILITY:
Inclusion Criteria:

1. The presence of written informed consent of the patient to participate in the study
2. Availability of examination data allowing for the verification or exclusion of cardiac and cardiac-associated pathology
3. Age 18 years old and older

Non-inclusion criteria:

1. Patients with an implanted permanent pacemaker;
2. ECG changes that prevent spectral analysis;
3. Conditions that may impair the quality of the ECG recording (Parkinson's disease, essential tremor, etc.);
4. Conditions that make ECG recording in lead I impossible (congenital anomalies of the upper limbs, traumatic amputation of the upper limbs).
5. Lack of written informed consent from the patient to participate in the study.

Exclusion Criteria:

1. Poor quality of the ECG recording on a single-channel ECG monitor
2. Insufficient examination data to verify or exclude cardiac or cardiac-associated pathology;
3. Patient's unwillingness to continue participating in the study for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with or without cardiac and cardiac-associated pathologies over 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-05-13 (Estimated)

PRIMARY OUTCOMES:
Parameters of single-channel ECG that significantly correlate with the presence of various cardiac and cardiac-associated pathologies | through study completion, an average of 2 years
  comparison of the presence of cardiac and cardiac-associated pathology by the results of full examination (laboratory, clinical and instrumental) with the results of the presence of valvular heart defects obtained using the mathematical model of a single-channel ECG monitor
Determination of sensitivity of various cardiac and cardiac-associated pathologies of multivariate models for analyzing single-channel electrocardiogram data | through study completion, an average of 2 years
  comparison of the presence of cardiac and cardiac-associated pathology by the results of full examination (laboratory, clinical and instrumental) with the results of the presence of valvular heart defects obtained using the mathematical model of a single-channel ECG monitor
Determination of specificity of various cardiac and cardiac-associated pathologies of multivariate models for analyzing single-channel electrocardiogram data | through study completion, an average of 2 years
  comparison of the presence of cardiac and cardiac-associated pathology by the results of full examination (laboratory, clinical and instrumental) with the results of the presence of valvular heart defects obtained using the mathematical model of a single-channel ECG monitor
Determination of diagnostic accuracy of various cardiac and cardiac-associated pathologies of multivariate models for analyzing single-channel electrocardiogram data | through study completion, an average of 2 years
  comparison of the presence of cardiac and cardiac-associated pathology by the results of full examination (laboratory, clinical and instrumental) with the results of the presence of valvular heart defects obtained using the mathematical model of a single-channel ECG monitor

IPD SHARING:
Plan to Share IPD: No
It is not possible to provide documentation due to the prohibition received from the local ethics committee

REFERENCES:
- [Background] A screening method for predicting left ventricular dysfunction based on spectral analysis of a single-channel electrocardiogram using machine learning algorithms / N. Kuznetsova, Zh. Sagirova, A. Suvorov [et al.] // Biomedical Signal Processing and Control. - 2023. - Vol. 86. - P. 105219. - DOI 10.1016/j.bspc.2023.105219. - EDN APQSQF.
- [Background] Complex automated remote system for assessing hemodynamic parameters when analyzing the native signal of a single-channel ECG and pulse wave using machine learning techniques / N. O. Kuznetsova, Zh. N. Sagirova, E. A. Sultygova [et al.] // Russian Journal of Cardiology. - 2023. - T. 28, No. S7. - pp. 41-42. - EDN LZGDKG.
- [Background] A Systematic Review on the Effectiveness of Machine Learning in the Detection of Atrial Fibrillation / A. L. Wuraola, B. Al-Dwa, D. Shchekochikhin [et al.] // Current Cardiology Reviews. - 2024. - Vol. 20. - DOI 10.2174/011573403x293703240715104503. - EDN XQZPAY.
- [Background] A single-lead ECG based cardiotoxicity detection in patients on polychemotherapy / D. F. Mesitskaya, Z. Z. A. Fashafsha, M. G. Poltavskaya [et al.] // IJC Heart and Vasculature. - 2024. - Vol. 50. - P. 101336. - DOI 10.1016/j.ijcha.2024.101336. - EDN XMKKZY.
- [Background] Kuznetsova N.O., Alekseeva A.M., Mamedzade F.E., Sedov V.P., Kopylov F.Yu., Syrkin A.L., Chomakhidze P.Sh. Screening for heart defects when analyzing an electrocardiogram using machine learning methods (literature review) // Bulletin of new medical technologies. Electronic edition. 2025. No. 1. Publication 1-6. DOI: 10.24412/2075-4094-2025-1-1-6. EDN KNFSNS
- [Background] Kuznetsova N.O., Nartova A.A., Kurbanalieva N.K., Adueva D.Sh., Chursina E.Yu., Zhvania R.E., Ustinova D.I., Kostikova A.S., Kazakova M.V., Tarnaeva L.A., Chomakhidze P.Sh., Kopylov F.Yu. Results of screening for heart rhythm disturbances using a single-channel electrocardiogram without the participation of medical personnel // Bulletin of new medical technologies. 2025. No. 1. P. 56-60. DOI: 10.24412/1609-2163-2025-1-56-60. EDN YWJLFH.
- See also: A single-channel ECG using machine learning techniques presentation — https://www.sechenov.ru/pressroom/news/v-sechenovskom-universitete-sostoitsya-v-mezhdunarodnyy-sammit-tsifroaytimed/?sphrase_id=3042055